CLINICAL TRIAL: NCT05145465
Title: Double Blinded Randomized Controlled Trial , Investigating the Efficacy of Telerehabilitation, Type 2 Diabetes Telerehabilitation,
Brief Title: The Effect of a Supervised Home-based Tele-rehabilitation Program on Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Garyfallia Pepera, Assistant Professor in Cardiovascular Physiotherapy/Cardiac Rehabilitation, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 716/23-09-2021
Record Dates: First submitted 2021-11-21; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 2; Telerehabilitation
Keywords: Supervised Exercise; Functional capacity; Hand grip
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Participants will undertake the first training session in the University of Thessaly under the supervision of a specialized physiotherapist in order to precept the exercises. All the other sessions will proceed via telerehabilitation program at their home. Participants will undergo an exercise home based program 3 times/week.
  The program will start with 10 minutes warm up exercise , 20 minutes continuous aerobic exercise ( 60-80% of target heart rate), 20 minutes resistance training exercise ( 30-50% 1RM), 5 minutes cool down and breathing exercises. For their safety patients will monitor glucose, blood pressure, pulse-oxygen and heart rate via, blood pressure monitor, pulse oximeter and smart-watch devices. They will be assessed at the beginning of the study and after the intervention ( at 6 weeks)
  Interventions: Other: Telerehabilitation group
- control group (No Intervention): The participants in this group will just receive the education session and they will continue their current medical therapies.They will be assessed at the beginning of the study and after the intervention ( at 6 weeks).

INTERVENTIONS:
Other: Telerehabilitation group — All the subjects in the telerehabilitation group will measure their heart rate and SpO2 with a pulse oximeter and blood pressure with digital sphygmomanometer themselves before ,during and after the end of each session for safety after they had been taught by physiotherapist. The patients will also oversee their blood sugar level before and after each session in order to prevent hypoglucemia events.
  The target heart rate for each patient will set at 60-80% of heart rate reserve plus the heart rate rest and wiil be calculated by the physiotherapist for each patient based on if they receive beta blockers medication or not.
  Arms: Telerehabilitation group

SUMMARY:
Tele-rehabilitation (TR) which carries health services distant through using electronic communication systems is an important treatment option. Although TR studies in musculoskeletal system, neurologic and cardio-pulmonary diseases are effective TR studies in type 2 DM patients are limited. TR interventions in patients with type 2 diabetes has not yet sufficiently defined and more studies with different exercise protocols will be an important step for the clinical value of this intervention but also for it's application in clinical practice.

Objective: The aim of this study is to evaluate the effectiveness of a telerehabilitation program on glucose control, functional capacity, muscle strength and quality of life in patients with type 2 diabetes.

Study design: It is a supervised-double blind randomized controlled trial, comparing two groups (a control group and a telerehabilitation group). The duration of the intervention will last 6 weeks.

Setting: home-based patients environments , only the first session in University of Thessaly for educational reason

Participants: A total of 22 patients with type 2 diabetes, regardless sex, aged 40 years and older will randomly assign to a telerehabilitation group (n = 11) and a control group (n = 11).

Measurements /Assessments Study data will be collected at baseline and after the intervention period ( 6 weeks) by two blinded physiotherapists, in University of Thessaly).

DETAILED DESCRIPTION:
Procedure:

The intervention program will last for 6 weeks and the patients in telerehabilitation-group will receive home based exercise program (by video-call with the supervision of a physiotherapist), 3 times per week and the total duration of each session will last for 60 minutes.

The control group will not receive any exercise intervention during that period but only an educational session.

Clinical assessments wiil be conducted before and 6 weeks after intervention and will include:

1. Functional capacity assesment tool : six minutes walking test ( 6MWT)
2. Physical activity] assesment tool : International Physical Activity Questionnaire (IPAQ).
3. Quality of life assesment tool : 36-Item Short Form Survey (SF-36) sf36
4. Hand grip strength assesment tool : Jamar Hydraulic Hand Dynamometer
5. Leg strength and endurance assesment tool 30 second chair stand test
6. Weight, hip , waist and BMI measurements
7. HbA1c level assesment tool : blood test

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2
* regulated blood sugar
* treatment by doctor
* greek language

Exclusion Criteria:

* no internet connection
* diabetes type 1
* recently surgery
* mental health problems

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 6 weeks
  The 6-min walk (6MW) test is commonly used to assess exercise capacity in patients and to track functional change resulting from disease progression or therapeutic intervention.
Physical activity | 6 weeks
  International Physical Activity Questionnaire - Short Form This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Hand grip strength | 6 weeks
  Jamar Hydraulic Hand Dynamometer The Jamar Hydraulic Hand Dynamometer can be used to measure isometric force and peak strength with five adjustable grip positions. The handle easily adjusts from 1 3/8" - 3 3/8" in half-inch increments. This helps track strength and rehabilitation over time.
Leg strength and endurance | 6 weeks
  30 second chair stand test Equipment: A chair with a straight back without arm rests (seat 17" high), and a stopwatch and count the number of times the patient comes to a full standing position in 30 seconds.
Quality of life (QOL) | 6 weeks
  36-Item Short Form Survey (SF-36) The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
HbA1c | 6 weeks
  HbA1c test, also known as the haemoglobin A1c or glycated haemoglobin test, is an important blood test that gives a good indication of how well your diabetes is being controlled
Body weight (kg) | 6 weeks
  Body weight will be calculated by a weighing scale and the unit of measurement will be in kilograms (kg)
Body height (cm) | 6 weeks
  Body height will be calculated by a stadiometer and the unit of measurement will be in centimeters (cm)
Hip size (cm) | 6 weeks
  hip measurements will be calculated by tape measure and the unit of measurement will be in centimeters ( cm)
Waist size (cm) | 6 weeks
  Waist measurements will be calculated by tape measure and the unit of measurement will be in centimeters ( cm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Greece